CLINICAL TRIAL: NCT02363361
Title: Treatment of Acute Cervical Spinal Cord Injury With Imatinib (Glivec®) - a Safety and Feasibility Study (EudraCT no 2014-002170-36)
Brief Title: Treatment of Cervical Spinal Cord Injury With Imatinib - a Safety and Feasibility Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Professor Mikael Svensson, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Professor Mikael Svensson, MD PhD, professor, MD, PhD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT no 2014-002170-36
Record Dates: First submitted 2015-02-03; First posted 2015-02-16 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Cervical Spinal Cord Injury
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imatinib (Experimental): Day 1. 800 mg, Day 2-14: 2 * 400 mg per day
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Day 1. 800 mg, Day 2-14: 2 * 400 mg per day
  Other Names: Glivec

SUMMARY:
This is a phase II, single center, open-label, non randomized clinical study to assess the uptake, safety and tolerability of Imatinib in acute Cervical Spinal Cord Injury patients. The aim is to determine if Imatinib reaches sufficient blood levels when given to patients with cervical spinal cord injury, via a gastric feeding tube, and also evaluate the safety and tolerability of this drug treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-80 years
2. Clinical signs of cervical spinal cord injury due to trauma.
3. In otherwise good health condition as determined by past medical history, physical examination, laboratory tests and vital signs
4. Patient that is conscious and oriented x 4 (regarding date/time, localisation, situation and personal details), with higher level of consciousness, i.e. Glasgow Coma Scale > 14, and is assessed to be competent to give informed consent.

Exclusion Criteria:

1. Diabetes (type I and II)
2. Ongoing cancer treatment
3. Known allergy to study drug Imatinib or its excipients
4. On current therapy with drugs which may interfere with Imatinib, (e.g. paracetamol, ketoconazole, itraconazole, erythromycin, clarithromycin, dexamethasone, phenytoin, carbamazepine, rifampicin, phenobarbital, fosphenytoin, primidon, Hypericum perforatum).
5. Female subjects lactating or with positive pregnancy test
6. Known liver or kidney disease
7. Any relevant surgical or medical condition which in the opinion of the investigator may interfere with the conduct of the study or the scientific results. This includes hemorrhagic conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in levels of Imatinib in plasma and cytokines in serum day 1-3, 7, 10, 14, 16, 19 | Day 1-3, 7, 10, 14, 16, 19

SECONDARY OUTCOMES:
Adverse events | Day 1-19

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Svensson, Prof.MD.PhD, Principal Investigator — Karolinska University Hospital